CLINICAL TRIAL: NCT04338490
Title: Effect of a Visual Feedback Device in Cardiopulmonary Resuscitation Training in AHA Certified ACLS Courses: Randomized Clinical Trial
Brief Title: Effect of the Use of a Visual Feedback Device in RCP Trainings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Carina Trindade de Castro, Principal researcher, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5637/19
Record Dates: First submitted 2020-01-16; First posted 2020-04-08 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Simulation Training
Keywords: cardiopulmonary ressuscitattion; education medical continuing; emergency medical services; simulation training; feedback dummy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Device: Feedback mannequim
- Control (No Intervention)

INTERVENTIONS:
Device: Feedback mannequim — The intervention group received rcp training with their performance being evaluated in real time so that they could correct themselves
  Arms: Intervention

SUMMARY:
To verify the efficacy of manikins with feedback in the training of physicians and nurses in the courses of Advanced Cardiac Life Support (ACLS) authorized by the American Heart Association (AHA) when compared to the traditional training form.

DETAILED DESCRIPTION:
Introduction: The Cardiopulmonary Arrest (CRP) is the largest medical emergency, training is fundamental for a good performance in Cardiopulmonary Resuscitation (CPR). In a realistic simulation scenario, the results tend to improve with the use of feedback manikins that evaluate the quality parameters in CPR and show in real time what the rescuer needs to improve in order to be successful in training and increase the probability of success in future real care. Objective: To verify the efficacy of the manikins with feedback in the training of physicians and nurses in the courses of Advanced Cardiac Life Support (ACLS) authorized by the American Heart Association (AHA). Methods: Comparison of CPR performance of ACLS students. The intervention group will be submitted to the real-time feedback of the manikins, the control group will receive feedback from the instructor. Statistical analysis will consist of inter-group comparisons and will cover mean, standard deviation, and parametric tests such as Student's T test. The results will be related to the characteristics of the sample, including anthropometric profile, profession, training time, practice area, previous training with a focus on CPR and physical exercise practice.

ELIGIBILITY:
Inclusion Criteria: Be an ACLS student and sign the TCLE. -

Exclusion Criteria: Refusing to sign the TCLE

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
The feedback mannequim is as effective as an AHA instructor | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Juarez Dr Neuhaus Barbisan, Study Director — Instituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul - Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nolan JP, Soar J, Smith GB, Gwinnutt C, Parrott F, Power S, Harrison DA, Nixon E, Rowan K; National Cardiac Arrest Audit. Incidence and outcome of in-hospital cardiac arrest in the United Kingdom National Cardiac Arrest Audit. Resuscitation. 2014 Aug;85(8):987-92. doi: 10.1016/j.resuscitation.2014.04.002. Epub 2014 Apr 15. PMID 24746785
- [Background] Austin AL, Spalding CN, Landa KN, Myer BR, Cure D, Smith JE, Platt G, King HC. A Randomized Control Trial of Cardiopulmonary Feedback Devices and Their Impact on Infant Chest Compression Quality: A Simulation Study. Pediatr Emerg Care. 2020 Feb;36(2):e79-e84. doi: 10.1097/PEC.0000000000001312. PMID 29084067
- [Background] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995
- [Background] Choi B, Asselin N, Pettit CC, Dannecker M, Machan JT, Merck DL, Merck LH, Suner S, Williams KA, Jay GD, Kobayashi L. Simulation-based Randomized Comparative Assessment of Out-of-Hospital Cardiac Arrest Resuscitation Bundle Completion by Emergency Medical Service Teams Using Standard Life Support or an Experimental Automation-assisted Approach. Simul Healthc. 2016 Dec;11(6):365-375. doi: 10.1097/SIH.0000000000000178. PMID 27509064
- [Background] Iskrzycki L, Smereka J, Rodriguez-Nunez A, Barcala Furelos R, Abelarias Gomez C, Kaminska H, Wieczorek W, Szarpak L, Nadolny K, Galazkowski R, Ruetzler K, Ladny JR. The impact of the use of a CPRMeter monitor on quality of chest compressions: a prospective randomised trial, cross-simulation. Kardiol Pol. 2018;76(3):574-579. doi: 10.5603/KP.a2017.0255. Epub 2018 Jan 3. PMID 29297195
- [Background] Kirkbright S, Finn J, Tohira H, Bremner A, Jacobs I, Celenza A. Audiovisual feedback device use by health care professionals during CPR: a systematic review and meta-analysis of randomised and non-randomised trials. Resuscitation. 2014 Apr;85(4):460-71. doi: 10.1016/j.resuscitation.2013.12.012. Epub 2013 Dec 21. PMID 24361457
- See also: Simulation-based learning in continuing medical education: analysis of student and teacher perceptions of a Hospital in Rio de Janeiro — http://dx.doi.org/10.1590/S0100-55022014000400007